CLINICAL TRIAL: NCT01693614
Title: An Open-label Phase II Study of BKM120 in Subjects With Relapsed and Refractory Diffuse Large B-cell Lymphoma, Mantle Cell Lymphoma and Follicular Lymphoma
Brief Title: Safety and Efficacy of BKM120 in Relapsed and Refractory NHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120Z2402; 2012-002208-41
Record Dates: First submitted 2012-09-04; First posted 2012-09-26 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Diffuse Large B-cell Lymphoma, Mantle Cell Lymphoma, Follicular Lymphoma
Keywords: Diffuse large B-cell lymphoma, Mantle cell lymphoma, Follicular lymphoma, PI3K inhibitor, Non-Hodgkin lymphoma, NHL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DLBCL Cohort (Experimental): Diffuse large B-cell lymphoma cohort
  Interventions: Drug: Buparlisib
- MCL Cohort (Experimental): Mantle cell lymphoma cohort
  Interventions: Drug: Buparlisib
- FL Cohort (Experimental): Follicular lymphoma cohort
  Interventions: Drug: Buparlisib

INTERVENTIONS:
Drug: Buparlisib — 100 mg hard gelatin capsules administered orally, once daily in cycles of 28 days
  Other Names: BKM120

SUMMARY:
This is a phase II study evaluating the safety, tolerability and efficacy of BKM120 in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL), mantle cell lymphoma (MCL) or follicular lymphoma (FL).

ELIGIBILITY:
Inclusion Criteria:

1. Patient had a histologically confirmed diagnosis of mantle cell lymphoma, follicular lymphoma, or diffuse large B cell lymphoma.
2. Patient had relapsed or refractory disease and received at least one prior therapy.
3. Patient with diffuse large B cell lymphoma had received or was ineligible for autologous or allogeneic stem cell transplant.
4. Patient had at least one measurable nodal lesion (≥2 cm) according to Cheson criteria (Cheson 2007). In case where the patient had no measurable nodal lesions ≥ 2 cm in the long axis at baseline, then the patient must have had at least one measurable extra-nodal lesion.
5. Patient had an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Patient had adequate bone marrow and organ function.

Exclusion Criteria:

1. Patient had received previous treatment with PI3K inhibitors
2. Patient had evidence of graft versus host disease (GVHD).
3. Patient had active or history of central nervous system (CNS) disease.
4. Patient had a concurrent malignancy or had a malignancy within 3 years of study enrollment (with the exception of adequately treated basal or squamous cell carcinoma or non-melanomatous skin cancer).
5. Patient had a score ≥ 12 on the PHQ-9 questionnaire.
6. Patient had a GAD-7 mood scale score ≥ 15.
7. Pregnant or nursing women
8. Patient who did not use highly effective contraception methods to avoid becoming pregnant or conceiving offspring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center Univ Nebraska, Omaha, Nebraska
  - Memorial Sloan Kettering Dept of Onc., New York, New York
  - Medical University of South Carolina -Hollings Cancer Center Medical Univ of South Carolina, Charleston, South Carolina
  - University of Texas MD Anderson Cancer Center Dept.ofMDAndersonCancerCtr(3), Houston, Texas
- Belgium (2):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Yvoir
- France (3):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Rennes
- Germany (2):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Milan, MI, Italy
- South Korea (2):
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Korea
- Spain (2):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Samsun

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Younes A, Salles G, Martinelli G, Bociek RG, Barrigon DC, Barca EG, Turgut M, Gerecitano J, Kong O, Pisal CB, Tavorath R, Kim WS. Pan-phosphatidylinositol 3-kinase inhibition with buparlisib in patients with relapsed or refractory non-Hodgkin lymphoma. Haematologica. 2017 Dec;102(12):2104-2112. doi: 10.3324/haematol.2017.169656. Epub 2017 Sep 29. PMID 28971900

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Primary reason for not completing is presented
Period: Overall Study
Arm/Group | DLBCL Cohort | MCL Cohort | FL Cohort
Started | 26 | 22 | 24
Completed | 0 | 0 | 0
Not Completed | 26 | 22 | 24
Not completed — Adverse Event | 7 | 11 | 5
Not completed — Disease progression | 11 | 8 | 7
Not completed — Protocol Violation | 5 | 2 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 4
Not completed — Withdrawal by subject/guardian | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DLBCL Cohort | MCL Cohort | FL Cohort | Total
Number analyzed (Participants) | 26 | 22 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (14.57) | 67.9 (8.56) | 61.4 (13.11) | 62.9 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 11 | 23
  Male | 18 | 18 | 13 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 19 | 17 | 21 | 57
  Black | 0 | 0 | 1 | 1
  Asian | 3 | 2 | 2 | 7
  Other | 4 | 3 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) and Disease Control Rate (DCR) Per Investigator at 6 Months (FAS)
Description: Overall Response rate is the percentage of patients in a cohort who experienced either complete response (CR) or partial response (PR) during their follow-up after treatment start divided by the total percentage of patients included in the corresponding cohort according to Cheson criteria The analysis for each cohort was based on an exact binomial test comparing the ORR to the reference level of 10% (null hypothesis) in the FAS. The test for each cohort used a significance level of 5%. The ORR was presented together with an exact 95% Clopper- Pearson confidence interval. Disease Control Rate (DCR progressive. Disease Control Rate (DCR) was the percentage of patients with CR, PR or SD (stable disease). Patients for whom the best response after treatment start was missing, unknown (UNK) or progressive disease (PD) were considered non-responders and were counted in the denominator for the estimation of the ORR
Time Frame: Baseline up to 6 months
Population: different numbers represents satisfying particular criteria
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DLBCL Cohort | MCL Cohort | FL Cohort
Number analyzed (Participants) | 26 | 22 | 24
percentage of participants
  ORR | 11.5 [2.45 to 30.15] | 22.7 [7.82 to 45.37] | 25.0 [9.77 to 46.71]
  DCR | 30.8 [14.33 to 51.79] | 81.8 [59.72 to 94.81] | 87.5 [67.64 to 97.34]

2. Secondary Outcome: Progression- Free Survival (PFS) Based on Investigator Assessment (FAS)
Description: Progression-free survival (PFS) is the time from the date of treatment start to the date of the first documented progressive disease (PD) or death due to any cause using Kaplan-Meier method by cohort.
Time Frame: Baseline up to approximately 44 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DLBCL Cohort | MCL Cohort | FL Cohort
Number analyzed (Participants) | 26 | 22 | 24
months | 1.8 [1.51 to 4.01] | 11.3 [3.81 to 38.90] | 9.1 [3.75 to 14.46]

3. Secondary Outcome: Duration of Response for Diffuse Large B-cell Lymphoma (DLBCL), and Follicular Lymphoma (FL) Cohorts (FAS)
Description: Duration of response is the time from the date of first occurrence of complete response (CR) or partial response (PR) to the date of the first documented progressive disease (PD) or death due to any cause
Time Frame: Baseline up to approximately 18 months
Population: Number analyzed represents participants satisfying criteria for duration of response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DLBCL Cohort | FL Cohort
Number analyzed (Participants) | 3 | 6
months | 2.2 [1.15 to NA] — Not able to estimate due to insufficient number of participants with events | 11.0 [3.94 to NA] — Not able to estimate due to insufficient number of participants with events

4. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With OS Events (FAS)
Description: Overall survival (OS) is the time from treatment start to the date of death due to any cause. Participants not known to have died were censored at the date of their last visit
Time Frame: Baseline up to approximately 44 months
Measure: Number; unit: percentage of participants
Arm/Group | DLBCL Cohort | MCL Cohort | FL Cohort
Number analyzed (Participants) | 26 | 22 | 24
percentage of participants
  OS events | 50.0 | 22.7 | 8.3
  Number censored | 50.0 | 77.3 | 91.7

5. Secondary Outcome: Percentage of Participants - Overall Survival- Kaplan Meier Estimates (FAS)
Description: Overall survival (OS) is the time from treatment start to the date of death due to any cause. Estimates done by cohort using Kaplan-Meier method with 95% confidence intervals
Time Frame: Baseline up to approximately 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DLBCL Cohort | MCL Cohort | FL Cohort
Number analyzed (Participants) | 26 | 22 | 24
percentage of participants
  2 month | 83.6 [61.98 to 93.52] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  4 month | 66.9 [44.54 to 81.88] | 90.2 [66.23 to 97.47] | 100.0 [100.0 to 100.0]
  6 month | 43.8 [23.26 to 62.64] | 90.2 [66.23 to 97.47] | 95.2 [70.72 to 99.32]
  12 month | 43.8 [23.26 to 62.64] | 77.8 [50.38 to 91.25] | 95.2 [70.72 to 99.32]
  18 month | 43.8 [23.26 to 62.64] | 70.1 [41.09 to 86.73] | 95.2 [70.72 to 99.32]

6. Secondary Outcome: Overall Survival - Median (FAS)
Description: as for outcome 5
Time Frame: Baseline up approximately 44 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DLBCL Cohort | MCL Cohort | FL Cohort
Number analyzed (Participants) | 26 | 22 | 24
months | 5.2 [3.06 to NA] — Not able to estimate due to insufficient number of participants with events | NA [15.64 to NA] — Not able to estimate due to insufficient number of participants with events | NA [22.74 to NA] — Not able to estimate due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 18 months
Groups:
- DLBCL Cohort: DLBCL
- MCL Cohort: MCL
- FL Cohort: FL
Arm/Group | DLBCL Cohort | MCL Cohort | FL Cohort
All-Cause Mortality (participants affected / at risk) | 7/26 | 1/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 12/26 | 12/22 | 7/24
Other Adverse Events (participants affected / at risk) | 25/26 | 22/22 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DLBCL Cohort (N=26) | MCL Cohort (N=22) | FL Cohort (N=24)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Performance status decreased (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Meningitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Essential tremor (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 2 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DLBCL Cohort (N=26) | MCL Cohort (N=22) | FL Cohort (N=24)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 2
Cataract (Eye disorders) | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 9
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 8 | 6 | 10
Vomiting (Gastrointestinal disorders) | 3 | 0 | 3
Asthenia (General disorders) | 3 | 5 | 4
Face oedema (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 6 | 8 | 13
Oedema peripheral (General disorders) | 0 | 0 | 3
Pyrexia (General disorders) | 3 | 2 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 3
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 1
Weight decreased (Investigations) | 3 | 8 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 10 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 5
Memory impairment (Nervous system disorders) | 0 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 1
Tremor (Nervous system disorders) | 1 | 4 | 2
Agitation (Psychiatric disorders) | 1 | 3 | 1
Anxiety (Psychiatric disorders) | 6 | 7 | 5
Confusional state (Psychiatric disorders) | 0 | 2 | 1
Depression (Psychiatric disorders) | 8 | 7 | 6
Insomnia (Psychiatric disorders) | 2 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 4
Hypertension (Vascular disorders) | 0 | 4 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT01693614/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT01693614/SAP_001.pdf